CLINICAL TRIAL: NCT02997748
Title: Remote Ischemic Preconditioning to Prevent Acute Kidney Injury in High Risk Patients After Cardiac Surgery (RIPCRenal)
Brief Title: Remote Ischemic Preconditioning After Cardiac Surgery
Acronym: RIPCRenal
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Muenster (Other)
Collaborators: Else Kröner Fresenius Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 04-AnIt-16
Record Dates: First submitted 2016-12-15; First posted 2016-12-20 (Estimated); Last update posted 2018-01-30 (Actual); Status verified 2018-01

CONDITIONS: Cardiac Surgery, Aortocoronary Bypass
Keywords: acute kidney injury; cardiac surgery; Remote ischemic preconditioning; [TIMP-2]*[IGFBP7]
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Observational group (No Intervention): No intervention, standard care
- Sham RIPC (Sham Comparator): Three cycles of 5- min upper limb sham ischemia
  Interventions: Procedure: Remote ischemic preconditioning (RIPC)
- RIPC-Group 1 (Experimental): Three cycles of 5- min upper limb ischemia
  Interventions: Procedure: Remote ischemic preconditioning (RIPC)
- RIPC-Group 2 (Experimental): Three cycles of 7-min upper limb ischemia
  Interventions: Procedure: Remote ischemic preconditioning (RIPC)
- RIPC-Group 3 (Experimental): Three cycles of 10-min upper limb ischemia
  Interventions: Procedure: Remote ischemic preconditioning (RIPC)
- RIPC-Group 4 (Experimental): Three Cycles of 5-min upper limb ischemia. If there is no response this will be followed by 2 cycles of 10-min upper-limb ischemia
  Interventions: Procedure: Remote ischemic preconditioning (RIPC)

INTERVENTIONS:
Procedure: Remote ischemic preconditioning (RIPC) — 3 cycles or more cycles of 5 to 10-min inflation of a blood-pressure cuff to 200 mm HG (or at least to a pressure 50 mmHG higher than the systolic arterial pressure) to one upper arm followed by 5 min reperfusion with the cuff deflated. In Non-Responder two additional cycles of 10 min cuff inflation will be performed in arm 6.
  Arms: RIPC-Group 1; RIPC-Group 2; RIPC-Group 3; RIPC-Group 4; Sham RIPC

SUMMARY:
Acute kidney injury (AKI) is a well-recognized complication after cardiac surgery with cardiopulmonary bypass (CPB). The aim of this study is to reduce the incidence of AKI by implementing remote ischemic preconditioning and to evaluate the dose-response relationship using the biomarkers urinary [TIMP-2] *[IGFBP7] in high risk patients undergoing cardiac surgery.

DETAILED DESCRIPTION:
Acute kidney injury (AKI) complicates 7-19% of cardiac surgical procedures. The investigators recently found that remote ischemic preconditioning (RIPC) using transient external compression of the upper arm prior to cardiac surgery was effective for reducing the occurrence of AKI (37.5% compared to 52.5% with sham; absolute risk reduction (ARR),15%; 95% CI, 2.56% to 27.44%; P=0.02). Fewer patients treated with RIPC received renal replacement therapy (RRT) (5.8% versus 15.8%; ARR, 10%; 95% CI, 2.25% to 17.75%; P=0.01). Moreover, the investigators found that the effectiveness of this intervention was strongly associated with the release of cell-cycle arrest biomarkers into the urine. Patients with urinary tissue inhibitor of metalloproteinases-2 and insulin-like growth factor-binding protein 7 ([TIMP-2]•[IGFBP7]) ≥ 0.5 (ng/ml)(ng/ml)/1000 before surgery had a significantly reduced rate of AKI compared to patients with lower urinary [TIMP-2]•[IGFBP7] concentration (relative risk (RR), 67%; 95% CI, 53% to 83%, P<0.001) whereas the biomarker concentrations after surgery predicted AKI as previously shown. This effect makes sense because cell-cycle arrest is thought to be part of the protective mechanisms endothelial cells use when exposed to stress. Stimulating these responses with RIPC should reduce AKI. Importantly, only 56% of patients treated with RIPC achieved an increase in urine [TIMP-2]•[IGFBP7] to ≥ 0.5, and only in this group was the intervention effective-patients that did not achieve this level showed no benefit.

Our goal is to eventually design and conduct a Bayesian 2-stage adaptive design sequence trial to evaluate the effectiveness of RIPC to prevent AKI in patients undergoing cardiac surgery. The dimensions of dose include duration, intensity and number of cycles. However, before this trial can be designed we need to answer 4 questions: i. Do baseline urinary [TIMP-2]•[IGFBP7] levels predict AKI (enrichment)? ii. Do [TIMP-2]•[IGFBP7] changes elicited by RIPC predict protection (RIPC efficacy measure)? iii. Is there a dose-response relationship between RIPC "dose" and [TIMP-2]•[IGFBP7]? iv. Is a dose-escalation RIPC protocol where doses are increased for non-responders, feasible and safe within the anesthesia workflow for cardiac surgery cases (practical)?

ELIGIBILITY:
Inclusion Criteria:

* Patients who are scheduled to undergo cardiac surgery with cardiopulmonary bypass
* Cleveland Clinic Score >=6

Exclusion Criteria:

* Acute myocardial infarction up to 7 days before surgery
* Age < 18 years
* Off-pump cardiac surgery
* Preexisting AKI
* Chronic kidney disease (GFR < 30 ml/min)
* Kidney transplantation within the last 12 months
* Peripheral arterial occlusive disease
* Pregnancy
* Hepatorenal syndrome
* Sulfonamide or thiazide medication within the last 7 days
* Participation in another interventional trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2016-12; Primary Completion 2019-06 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Change in urinary [TIMP-2]*[IGFBP7] | within 12 hours after CPB
  Biomarkers will be measured at different time points after to evaluate the effect of RIPC on [TIMP-2]*[IGFBP7]

SECONDARY OUTCOMES:
AKI within 72 hours | 72 h
Dialysis within 7 days of surgery | 7 days
All-cause-mortality at 90 days | 90 d
Dialysis at day 90 | 90 days
Renal recovery at day 90 | 90 days
MAKE 90 | 90 days
  major adverse kidney events

CONTACTS AND LOCATIONS:
Overall Officials: Melanie Meersch, Study Chair — University Hospital Muenster
Locations (1):
- University Hospital Muenster, Münster, Germany

IPD SHARING:
Plan to Share IPD: No